CLINICAL TRIAL: NCT01078519
Title: Combined Spinal and Epidural Anesthesia and Maternal Intrapartum Temperature During Vaginal Delivery: a Randomized Clinical Trial
Brief Title: Combined Anesthesia for Labor and Maternal Temperature
Acronym: feveranalg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Flavia Augusta de Orange, Instituto Materno infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCT00992524
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2007-12

CONDITIONS: Pyrexia; Abdominal Delivery
Keywords: Fever; anesthesia; Labor
MeSH Terms: conditions — Fever | interventions — Anesthesia, Spinal; Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massages baths (No Intervention): doulas, massages and baths
- Combined spinal-epidural anesthesia (Active Comparator): local anesthetics in low doses with opioids
  Interventions: Drug: Combined epidural and spinal anesthesia

INTERVENTIONS:
Drug: Combined epidural and spinal anesthesia — Obstetrics patients will relieve spinal anesthesia with local anesthesics and opioids associated with epidural anesthesia with local anesthetics in low concentrations with opioids
  Other Names: Local anesthetics; spinal opioides
  Arms: Combined spinal-epidural anesthesia

SUMMARY:
Maternal intra-partum fever commonly complicates the process of labour. Its occurrence is often regarded as being synonymous with the presence of chorioamnionitis. This inevitably results in the administration of antibiotics to the affected mother. Review of the literature however suggests that this approach is not always appropriate. Non-infective causes of this condition that are often overlooked include the use of epidural analgesia for pain relief, normal thermal physiological changes in women not using any form of analgesia and delivery in an overheated room. Women with certain risk factors such as nulliparity and a long latent phase of labour are also more prone to developing maternal intra-partum fever. Irrespective of its aetiology, maternal intra-partum fever carries risks both for the mother and her unborn child. Putting more thought into the care of these patients will go a long way in reducing the maternal and neonatal morbidity associated with this complication.The combined spinal-epidural (CSE) technique has been introduced in an attempt to reduce these adverse effects. CSE is believed to during labour provide more rapid onset of analgesia than epidural analgesia, The incidence of fever is significantly lower with CSE technique.

DETAILED DESCRIPTION:
The objective this study is determine the fever maternal incidence with CSE technique for labor analgesia.

METHODS: a randomized open clinical trial will be conducted involving Seventy healthy, term, nulliparous women in spontaneous labor were assigned to either CSE technique or non pharmacologic analgesia for labor.these patients will be randomly assigned to receive or not CSE technique for labor analgesia. Outcomes analysis wiil include maternal fever, pain intensity measured by visual analog scale, labor duration, c-section and instrumental delivery. statical analysis will performed using Mann-Whitney and Fisher" exact test 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* babies were presenting head first
* were expecting a vaginal delivery single fetal
* gestational age up to 37 weeks
* cervix length between 3-6 cm

Exclusion Criteria:

* Maternal fever before randomization
* Antibiotics before randomization
* haemostatic disorders during pregnancy
* severe preeclâmpsia-eclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Fever frequency | each hour
  We will measure the temperature each hour

SECONDARY OUTCOMES:
Incidence of c-section and instrumental delivery | within the delivery
  Will measure the instrumental delivery when the CSA technique is used

CONTACTS AND LOCATIONS:
Overall Officials: Flavia A Orange, Principal Investigator — IMIP